CLINICAL TRIAL: NCT02050932
Title: The Optimization of Iron Bioavailability of Supplements Using Hepcidin Levels in Humans: Effect of the Time of Administration and Consecutive Day Administration of Commonly Used Dosages
Brief Title: The Optimization of Iron Bioavailability of Supplements Using Hepcidin Levels in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EK 2013-N-41
Record Dates: First submitted 2013-11-08; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Iron Deficiency
Keywords: hepcidin; iron bioavailability; iron supplementation
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron absorption assessement (Experimental): 60 mg Fe as FeSO4 with stable isotopic labels participants will receive at different times of the day (total of three dosages) and follow a standardized diet scheme.
  Subjects will act as their own controls during the study
  Interventions: Dietary Supplement: 60 mg Fe as FeSO4 with stable isotopic labels

INTERVENTIONS:
Dietary Supplement: 60 mg Fe as FeSO4 with stable isotopic labels — Subjects will receive FeSo4 supplements labeled with stable isotopic labels (54Fe, 57Fe, 58Fe) and iron absorption will be measured for each administration

SUMMARY:
Background: Oral iron supplementation (OIS) is a widely-used strategy to treat iron deficiency anemia. However, absorption of OIS is often low and response is variable. To overcome this, large doses are given but this may reduce compliance due to gastric irritation. Thus, OIS doses should be low, while maximizing absorption. The prevailing serum hepcidin concentration (SHep) is the major determinant of iron absorption and erythrocyte iron utilization. Based on limited data in humans, SHep can be increased by a single OIS dose but the duration of the increase is uncertain: In a recent study conducted in our laboratory it has been found to last approx. 24 h. Also, there are few data on how the increase in SHep determines the absorption of further doses of oral iron. Is there a threshold SHep at which subsequent iron absorption is sharply reduced? Better understanding of this relationship would be valuable to design more effective and safer OIS regimens.

Objectives: 1) Determine whether two consecutive dosages of 60 mg Fe differently affect hepcidin response and iron bioavailability (Study 1) 2) Compare the bioavailability of iron supplement dosages given at different times of the day (Study 2).

Methods/Subjects: Healthy female subjects will be screened for low iron status. Anemic subjects will be excluded from the study. Thirty two subjects will be included with serum ferritin <20 µg/L, C-reactive protein <5 mg/L and Hemoglobin >117 g/L. Subjects will be randomized in two groups and their Hepcidin (sHep) and iron status markers monitored at day 1 (baseline). Subjects will receive iron supplement dosages of 60 mg with stable iron isotopes 54Fe, 57Fe, 58Fe in form of 4 mg of FeSO4. Prior administration blood samples will be collected to monitor sHep and iron status markers.

Outcome: The combined use of stable iron isotopes and a sensitive SHep assay will allow for better understanding of the iron-hepcidin relationship and this may enable design of more effective OIS regimens.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, no blood donation in the last 4 months, not pregnant, not lactating, not taking vitamin and mineral supplements 2 weeks prior the study, non smoker, weight <65 Kg, BMI between 18 and 25.
* No anemia (defined as 11.7 g/dl, Serum ferritin level < 20 microgram/L).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Iron absorption of stable isotopic tracers. | 14 days
  Stable iron isotopes will be administered under standardized conditions and close supervision. Iron absorption will be calculated from the shift in the normal isotopic abundance in Red blood cells 14 days after test meal incorporation.

SECONDARY OUTCOMES:
Iron status | 14 days
  To characterize participants, iron status will be assessed by measuring serum ferritin.
Inflammatory status | 14 days
  To characterize subjects participating to the study, C- reactive protein will be measured as inflammatory marker.
Hepcidin level | 14 days
  As a determinant of iron absorption (primary outcome) hepcidin level will be measured at all timepoint prior administration of stable isotopic label tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — ETH Zürich, Laboratory of Human Nutrition
Locations (1):
- ETH Zürich, Laboratory of Human Nutrition, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Moretti D, Goede JS, Zeder C, Jiskra M, Chatzinakou V, Tjalsma H, Melse-Boonstra A, Brittenham G, Swinkels DW, Zimmermann MB. Oral iron supplements increase hepcidin and decrease iron absorption from daily or twice-daily doses in iron-depleted young women. Blood. 2015 Oct 22;126(17):1981-9. doi: 10.1182/blood-2015-05-642223. Epub 2015 Aug 19. PMID 26289639